CLINICAL TRIAL: NCT04378686
Title: A Comparative Study of Symptom-driven Surveillance vs. Cross-sectional Serological Screening of SARS-CoV-2 Infection of Patients With End-stage Kidney Disease Receiving Renal Replacement Therapy
Brief Title: Serological Testing for COVID-19 (SARS-CoV-2) in ESKD
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S64000
Record Dates: First submitted 2020-05-05; First posted 2020-05-07 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: SARS-CoV 2; End Stage Renal Failure on Dialysis
Keywords: nasopharyngeal swab; Chest CT; serology
MeSH Terms: interventions — Dialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ESKD: Patients with ESKD and on treatment with any form of dialysis
  Interventions: Other: dialysis

INTERVENTIONS:
Other: dialysis — treatment with dialysis. This can be hemodialysis, hemodiafiltration, peritoneal dialysis

SUMMARY:
Starting in late 2019, the world is facing a pandemic with the SARS-CoV-2 virus. Patients with end-stage kidney disease and on treatment with renal replacement therapy are high risk patients, as they are unable to maximize social distancing.

We plan to gather epidemiological data using two different diagnostic approaches. We will compare a symptom-driven screening, in combination with a nasopharyngeal swab plus computed tomography (clinical approach) against serological surveillance.

DETAILED DESCRIPTION:
In late 2019, a cluster of patients with unexplained pneumonia was linked to a novel beta-coronavirus, now known as severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) 1. The world health organization subsequently has coined this disease as COVID-19. By the time the scientific community was alerted, the epidemiological data suggested that the virus had already spread to other regions of mainland China, as well as foreign cities with close transport links to the original epicenter 2. The world initially answered by divergent responses. Two months on, we are experiencing a devastating pandemic with local outbreaks across all continents.

As more and more patients arrive at the hospitals, our focus is drawn to the acute and the important issues, treating large numbers of patients in grave condition. The surge in patients requiring medical care may overwhelm even the most sophisticated healthcare systems 3. The approach adopted by almost all nations is to 'flatten the curve', i.e. to reduce peak demand of healthcare resources 4. While individual countries follow different paths, the common denominator is to maximize social distancing. The main goal is to reduce the basic reproduction number (R0) as much as possible, to ideally less than 1.

An overview of the clinical characteristics of confirmed cases in China alerted the world that young age does not protect against infection 5. Disease severity, however, varies by age with more elderly people becoming seriously ill, and by underlying medical condition(s) 6. The impact on peak medical demand thus will be even greater if we succeed in maximizing social distancing of the most vulnerable and most frail patients, those who are more likely to become seriously ill.

This is, however, difficult for dialysis patients who cannot self-isolate and cannot avoid multiple contacts per week with health care workers and other patients. While isolating dialysis patients and health care workers with a suspected SARS-CoV-2 infection is important to limit transmission of the virus, these measures are insufficient to avoid transmission since it is estimated that asymptomatic or paucisymptomatic people play a major role in the spread of the virus. So far, epidemiological data in patients on IHD during an SARS-CoV-2 outbreak are limited. A single case-series of cases from China has been reported in prepublication. 37 out of 230 patients were infected with SARS-CoV-2, of which 6 died (crude mortality rate 16.2%). The authors suggest that not all of these died directly from the consequences of COVID-19. However, adjudication of cause of death might differ in future case series.

The current gold standard for the diagnosis of acute respiratory syndrome due to SARS-CoV-2 (COVID-19) is the detection of viral RNA in respiratory tract samples. The sensitivity of a negative PCR result is, however, not 100%. False-negatives can occur, especially when using nasopharyngeal swabs (positivity rate estimated at 54%-74%) due to sampling error and in patients with low viral loads, especially in patients who present at day 8 or later and mild cases. While a CT scan can be a valuable tool in patients with a suspicion of COVID-9, measurement of antibodies against SARS-CoV-2 is the only reliable way to estimate the prevalence of SARS-CoV-2 infection since patients can be pauci-symptomatic or asymptomatic.

A number questions remain regarding the use of antibodies for epidemiologic studies and to determine immunity. Can someone have a colonization with SARS-CoV-2 without developing IgG antibodies? In this case, would this person be protected against reinfection? Doctors of the University of Bonn recently reported on April 9th (H. Streeck et al.,data not yet published) that only 15% of a sample of 1.000 inhabitants of the small town Gangelt, a local hotspot in North Rhine Westphalia tested positive for IgG antibodies. These data suggest that even in severely affected regions the critical threshold for herd immunity might not have been reached. This means that there is a significant risk of new outbreaks, particularly after schools might reopen later (maybe in summer 2020, and in fall 2020).

Given that dialysis patients are at the same time potentially more vulnerable to SARS-CoV-2 infection, and cannot self-isolate, it is important to closely monitor this group of patients. A second benefit of this population is that it easily accessible for blood sampling, and close clinical follow-up is ensured.

The aim of this study is to determine the prevalence of patients who were infected with SARS-CoV-2 by measuring IgG antibodies at different time points.

Trial objectives The aim of the current study is to collect epidemiological data of the incidence of severe acute respiratory syndrome Corona Virus type 2 (SARS-CoV-2) infections patients with end-stage kidney disease in a Belgian Hospital setting.

The objective is to compare two means of detection of infection, one symptom-driven surveillance and a second based on cross-sectional serology.

Primary endpoints Positive serology for SARS-CoV-2 at census date(s)

Secondary endpoints Detection of SARS-CoV-2 infection by symptom-driven surveillance

Trial Design Cross-sectional and longitudinal observational study of prevalent patients with end-stage kidney disease

ELIGIBILITY:
Inclusion Criteria:

* Patients with end-stage kidney disease (ESKD) receiving renal replacement therapy
* Age 18 years or older
* Treated at University Hospitals Leuven, or Jessa Ziekenhuis Hasselt
* Providing informed consent

Exclusion Criteria:

* Refusal to provide informed consent
* Transfer to another dialysis unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with end-stage kidney disease (ESKD) receiving renal replacement therapy
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Antibodies against SARS-CoV-2 | one year
  serology to test for IgG and IgM antibodies against SARS-CoV-2

CONTACTS AND LOCATIONS:
Overall Officials: Bjorn Meijers, MD, PhD, Principal Investigator — UZ Leuven
Locations (3):
- Belgium (3):
  - Jessa Ziekenhuis, Hasselt, Limburg
  - Sint Trudo, Sint-Truiden, Limburg
  - University Hospitals Leuven, Leuven

IPD SHARING:
Plan to Share IPD: Undecided
undecided